CLINICAL TRIAL: NCT05632874
Title: The Effect of Relaxing Breathing Exercise Applied to Patients Before Bone Marrow Biopsy on Vital Signs, Pain and Anxiety Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Ahmet Kolip, Principal Investigator, Uskudar University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UskudarUniveristy
Record Dates: First submitted 2022-11-09; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Bone Marrow Cancer
Keywords: bone marrow biopsy; pain; breathing exercise; anxiety
MeSH Terms: conditions — Bone Marrow Neoplasms; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breathing Exercise (Experimental)
  Interventions: Behavioral: relaxing breathing exercise

INTERVENTIONS:
Behavioral: relaxing breathing exercise — "Kumbhaka Pranayama", "Sama Vritti Pranayama" and "box breathing" breathing techniques will be applied to the patients.

SUMMARY:
There is no study in the literature that determined the effect of relaxing breathing exercise applied to patients before the BMB procedure on vital signs, pain and anxiety levels.

The aim of this study is to determine the effect of relaxing breathing exercise applied to patients before bone marrow biopsy on vital signs, pain and anxiety levels.

hypotheses H1. Relaxing breathing exercise applied to the patients before the bone marrow biopsy procedure reduces the anxiety level of the patients compared to the control group.

H2. Relaxing breathing exercise applied to the patients before the bone marrow biopsy procedure reduces the pain level of the patients compared to the control group.

H3. Relaxing breathing exercise applied to the patients before the bone marrow biopsy procedure is effective on the respiratory rate of the patients compared to the control group.

H4. Relaxing breathing exercise applied to the patients before the bone marrow biopsy procedure is effective on the pulse rate of the patients compared to the control group.

H5. Relaxing breathing exercise applied to the patients before the bone marrow biopsy procedure is effective on the blood pressure of the patients compared to the control group.

ELIGIBILITY:
* Being between the ages of 18-65
* The fact that a bone marrow biopsy will be performed for the first time
* Absence of sedative, anxiolytic drug use
* Absence of a situation that would hinder communication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analouge Scale | up to 1 mounth
  After the application, the pain level of the patients is expected to be low.

CONTACTS AND LOCATIONS:
Locations (1):
- Uskudar Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes